CLINICAL TRIAL: NCT04080596
Title: A Single Dose, Open Label, Drug-drug Interaction Study to Investigate the Pharmacokinetics, Pharmadynamics and Safety of HMS5552 Administered Alone or in Combination With Itraconazole in Patients With Type 2 Diabetes Mellitus
Brief Title: DDI Study to Investigate the Impact of Itraconazole on the Pharmacokinetics of Dorzagliatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMM0107
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Dorzagliatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential arm (Experimental): Dorzagliatin administered alone on Day 1; after wash-out, intraconazole was administered from Day 8 to Day 15, with Dorzagliatin administered together on Day 11.
  Interventions: Drug: Dorzagliatin

INTERVENTIONS:
Drug: Dorzagliatin — GKA for T2DM currently under clinical development
  Other Names: HMS5552

SUMMARY:
The purpose of this study is to investigate the impact of itraconzaole on the pharmacokinetics of Dorzagliatin.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65
* Body weight ≥ 50 kg
* BMI ≥ 19.0 kg/m2 and ≤ 30.0 kg/m2
* HbA1c ≥ 7% and ≤ 10.5%
* FPG ≥ 7.5 mmol/L and ≤ 13.3 mmol/L

Exclusion Criteria:

* T1DM
* Use of prescription or OTC medications, and herbal within 14 days prior to dosing
* Blood donation
* Any surgery or treatment that may impact the ADME of the drug

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 96 hours
  Peak concentration
AUClast | up to 96 hours
  Area under the curve

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No